CLINICAL TRIAL: NCT06457620
Title: Comparison of Telerehabilitation vs Clinical Setup Rehabilitation in TKR Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/725
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy (Experimental)
  Interventions: Behavioral: Conventional Physiotherapy
- traditional physical treatment (Other)
  Interventions: Other: Traditional Physical Preatment

INTERVENTIONS:
Behavioral: Conventional Physiotherapy — Each participant received conventional physiotherapy at the clinic as a part of their management plan. Group A exercise was five times a week for thirty minutes, beginning on the third day after total knee arthroplasty (TKA). The program aimed to improve leg strength, core stability, balance, and overall performance through exercise instructions. The baseline evaluation was completed one day before the TKA, and the posttest was completed four weeks after the TKA.
  Arms: conventional physiotherapy
Other: Traditional Physical Preatment — Each participant got traditional physical treatment during a video conference as part of telerehabilitation. The physiotherapy assistant contacted Group B to arrange a virtual follow-up clinic appointment via Zoom or WhatsApp, along with a 4-week program. We inquired about the patient's level of satisfaction with their TKR procedure. The patient was informed that clinical photos were taken, and the video call was to be recorded. Before the virtual clinic, each patient's verbal agreement was acquired. With workout instructions, the program pursued to enhance leg strength, core stability, balance, and overall performance. The posttest was conducted four weeks after the TKA, and the baseline assessment was finished one day before the procedure.
  Arms: traditional physical treatment

SUMMARY:
This study examines the feasibility, attainability, and patient satisfaction of telerehabilitation and clinical consultation rehabilitation.

DETAILED DESCRIPTION:
The objective is to assess whether telerehabilitation can provide comparable or significantly better outcomes in terms of functional recovery, pain management, improved range of motion, and patient satisfaction for Total Knee Replacement (TKR) patients. If telehealth interventions prove successful, they can be implemented to increase access to high-quality rehabilitation treatments and enhance healthcare delivery. Evidence-based findings from this study can help healthcare providers make educated decisions about incorporating telerehabilitation into post-operative rehabilitation protocols, thereby enhancing patient care and optimizing resource utilization in orthopedic settings.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with TKR
* Older Age above 65
* Patient communicates with medical staff
* Patient with cemented TKA
* Patients who underwent TKA owing to degenerative arthritis

Exclusion Criteria:

* Older patients aged >75 years
* Patient with a history of knee joint surgery before TKA
* Patient who possibly had a systematic inflammatory disease such as rheumatoid arthritis.
* Patients with difficulty in seeing, hearing, and walking independently
* Patients having a history of mental illnesses (Stroke, Multiple sclerosis, Parkinsonism, Alzheimer's Disease)
* Patient history of severe mobility disorder
* Systemic illness (Liver Failure, Active cancer, Cardiopulmonary distress)

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WoMAC) | 12 Months
  The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. ,
Knee Outcome Survey-Activities of Daily Living (KOS-ADLS) | 12 months
  The Knee Outcome Survey (KOS) is a patient-completed questionnaire that provides a percentage of disability during every day activities (activities of daily living subscale) or sports (sports activity subscale). The lower the percentage, the higher the disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Acti Life Physiotherapy and Rehabilitation Center Horizon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No